CLINICAL TRIAL: NCT01261546
Title: MULTICENTRIC, PHASE II, CLINICAL TRIAL CORTICOIDS FOR EMPYEMA AND PLEURAL EFFUSION IN CHILDREN
Brief Title: Clinical Trial Corticoids For Empyema And Pleural Effusion In Children
Acronym: CORTEEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Infanta Sofia (Other)
Collaborators: Pediatrics Spanish Association (Madrid and Castilla-La Mancha Pediatric Association) (Unknown); Spanish Ministry of Health. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hospital Infanta Sofia; 2009-012963-33 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Parapneumonic Pleural Effusion; Empyema
Keywords: pleural effusion, empyema, corticoids, dexamethasone
MeSH Terms: conditions — Empyema; Pleural Effusion | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): * Dexamethasone 0,25mg/kg, IV, q.i.d. for 2 days.
  * Cefotaxime 200 mg/kg, IV, q.d. until discharge criteria are present
  * Ranitidine 5 mg/kg IV, q.d. for 2 days
  * Amoxicillin/Clavulanic acid orally (80mg/kg/day) during 15 days.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Normal saline 0,6 ml/kg, IV, q.i.d. for 2 days.
  * Cefotaxime 200 mg/kg, IV, q.d. until discharge criteria are present.
  * Ranitidine 5 mg/kg IV, q.d. for 2 days.
  * Amoxicillin- Clavulanic acid 80mg/kg p.o., q.d. during 15 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — * Dexamethasone 0,25mg/kg, IV, q.i.d. for 2 days.
  * Cefotaxime 200 mg/kg, IV, q.d. until discharge criteria are present
  * Ranitidine 5 mg/kg IV, q.d. for 2 days
  * Amoxicillin/Clavulanic acid orally (80mg/kg/day) during 15 days.
  Arms: Dexamethasone
Drug: Placebo — Normal saline 0,6 ml/kg, IV, q.i.d. for 2 days.
  * Cefotaxime 200 mg/kg, IV, q.d. until discharge criteria are present.
  * Ranitidine 5 mg/kg IV, q.d. for 2 days.
  * Amoxicillin- Clavulanic acid 80mg/kg p.o., q.d. during 15 days.
  Arms: Placebo

SUMMARY:
STUDY JUSTIFICATION

1. Scientific evidence of the usefulness of corticosteroid use for infectious diseases: Corticosteroids along with antibiotic use improve survival in some infectious processes provide long term benefits and improve symptoms in many others.
2. Clinical Observation: the investigators observed that patients with parapneumonic pleural effusion and associated bronchospasm who were treated with corticosteroids for their bronchospasm, evolved to healing before patients who were not treated with corticosteroids (average admission days 10 vs. 17).
3. Rationale: the anti-inflammatory effect has been the rationale for the use of dexamethasone as an inhibitor of the inflammatory response observed after the first dose of parenteral antibiotic in bacterial meningitis. A similar effect is likely to occur in pneumonia with pleural effusion. It can be therefore hypothesized that Dexamethasone could inhibit an excessive inflammatory response by mesothelial and inflammatory cells during the early phases of parapneumonic empyema, reducing its severity and hence its complications.

OBJECTIVES

1. Principal: to investigate if dexamethasone 0,25mg/kg q.i.d. added to standard antibiotic therapy reduces time to resolution of parapneumonic pleural effusion.
2. Secondary:

2.1. Evaluate the effect of dexamethasone 0,25mg/kg q.i.d. added to standard antibiotic therapy on the development of complications during pleural effusion episode.

2.2. Evaluate the incidence of severe and non severe adverse events associated with the new treatment versus standard therapy.

METHODS

1. Study design: exploratory (pilot), randomized, double blinded, placebo controlled, parallel stratified design, multicentric.
2. Participating Hospitals (n=56, 7 patients per center):

   * Hospital Infanta Sofía (S. Sebastián de los Reyes, Madrid).
   * Hospital Universitario de Getafe
   * Hospital Universitario Ramón y Cajal, Madrid.
   * Hospital Universitario Materno-Infantil Carlos Haya, Málaga.
   * Hospital Infantil La Paz, Madrid.
   * Hospital U. Gregorio Marañón
   * Hospital U. Príncipe de Asturias
   * Hospital Virgen de la Salud, Toledo
3. Endpoints:

   3.1. Primary: time to resolution. 3.2. Secondary endpoints:
   1. Effectiveness: number of children with complications.
   2. Safety (expected number: none). i) Hyperglycemia ii) Signs of gastrointestinal bleeding iii) Need of transfusion iv) Oropharyngeal Candidiasis v) Allergic reaction vi) Other adverse reactions described in the Medication Guide.
4. Treatment arms:

3.1. Control (0)

* Normal saline 0,6 ml/kg, IV, q.i.d. for 2 days.
* Cefotaxime 150 mg/kg, IV, q.d. until discharge criteria are present.
* Ranitidine 5 mg/kg IV, q.d. for 2 days.
* Amoxicillin- Clavulanic acid 80mg/kg p.o., q.d. during 15 days.

3.2. Study treatment: (1)

* dexamethasone 0,25mg/kg, IV, q.i.d. for 2 days.
* Cefotaxime 150 mg/kg, IV, q.d. until discharge criteria are present
* Ranitidine 5 mg/kg IV, q.d. for 2 days
* Amoxicillin/Clavulanic acid orally (80mg/kg/day) during 15 days.

  4. INCLUSION CRITERIA
* Patients between 1 and 14 year old.
* Presence of pneumonia diagnosed by clinical and radiographic criteria: cough, fever and radiological consolidation.
* Evidence of pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 1 and 14 year old.
* Presence of pneumonia diagnosed by clinical and radiographic criteria: cough, fever and radiological consolidation.
* Evidence of pleural effusion.

Exclusion Criteria:

* Allergy to any of the drugs included in the study.
* Immunodeficiency.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
time to resolution | 1 month after admission
  days from diagnosis until criteria for cure

SECONDARY OUTCOMES:
number of children with complications. | 3 months after diagnosis
  number of children with complications.
Number of children with complications attributable to corticoids | 3 months
  Hyperglycemia Signs of gastrointestinal bleeding Need of transfusion Oropharyngeal Candidiasis Allergic reaction

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Carlos Haya, Málaga, Andalusia
  - Complejo Hospitalario Toledo, Toledo, Castille-La Mancha
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Infantil La Paz, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid

REFERENCES:
- [Derived] Tagarro A, Otheo E, Baquero-Artigao F, Navarro ML, Velasco R, Ruiz M, Penin M, Moreno D, Rojo P, Madero R; CORTEEC Study Group. Dexamethasone for Parapneumonic Pleural Effusion: A Randomized, Double-Blind, Clinical Trial. J Pediatr. 2017 Jun;185:117-123.e6. doi: 10.1016/j.jpeds.2017.02.043. Epub 2017 Mar 28. PMID 28363363